CLINICAL TRIAL: NCT06585384
Title: Safety of a Strategy Combining Etanercept Administration with Repeated Contrast Ultrasound in Patients with Alzheimer's Disease: Phase I Study
Brief Title: Safety of a Strategy Combining Etanercept Administration with Repeated Contrast Ultrasound in Patients with Alzheimer's Disease
Acronym: BRAINWAVES
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPX_2023_4
Record Dates: First submitted 2024-07-31; First posted 2024-09-05 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- etanercept and repeated contrast ultrasound (Experimental)
  Interventions: Combination Product: etanercept and repeated contrast ultrasound

INTERVENTIONS:
Combination Product: etanercept and repeated contrast ultrasound — Strategy combining 9 weeks of etanercept administration (50mg/week) with 5 weeks of repeated contrast ultrasound of 2 sessions per day, 5 days per week (from the fifth week of etanercept treatment)

SUMMARY:
Alzheimer's disease (AD) is a clinico-pathological entity combining multiple and varied neuropathological lesions with characteristic abnormal accumulations (amyloid Beta (Aβ) plaques and neurofibrillary degeneration (NFD)), neuroinflammation, as well as neuronal and synaptic suffering.

To date, only symptomatic treatments are available, with no proven effect on neuropathological lesions or on the clinical course of the disease.

Anti-TNF alpha could be a therapeutic agent of choice in the treatment of central nervous sytem (CNS) diseases with an inflammatory component, such as AD. Unfortunately, their high molecular weight prevents them from passively crossing the blood brain barrier (BBB). In a pilot study published in 2006, etanercept was administered intrathecally to AD patients with encouraging clinical effects.

Transient opening of the tight junctions between the endothelial cells of the BBB by delivering High Intensity Focalised Ultrasounds (HIFU) in combination with an intravenous injection of microbubbles is a strategy that could improve bioavailability. Studies suggest that the oscillation of microbubbles in the ultrasound field generates microcurrents that induce shear forces responsible for a transient opening of the BBB. Ultrasound can be focused or unfocused and open the BBB diffusely or selectively over defined regions of the brain. This technique was first used to open the BBB in humans in 2001.

Transient opening of the BBB is also thought to modulate the immune response in the CNS, leading to a reduction in the intracerebral load of Aβ. In an Alzheimer's mouse model, several studies using ultrasound devices to open the BBB have shown a reduction in the intracerebral load of Aβ (up to 75%) and an improvement in the memory faculties and cognitive performance of the animals.

In humans, two clinical trials have assessed the safety of using ultrasound-assisted BBB disruption devices in AD patients. These were the Sonocloud® (Carthera) and ExAblate® (InSightec) devices. The Sonocloud® device is an extra-dural ultrasound emitter implanted under local anaesthetic. Enrolment was completed in October 2020, but the results of the trial are not yet available (NCT03119961). The phase I study on 5 patients evaluating the ExAblate® device coupled with the injection of gas microbubbles demonstrated reversible opening of the BBB with no serious adverse effects for the patients. No effect on intracerebral Aβ load or cognitive or behavioural improvement was demonstrated. The ExAblate® device is not implantable and is therefore less invasive than the Sonocloud® device. However, it requires MRI monitoring and the transducers used often generate high levels of heat, requiring the use of a water cooling system to avoid the risk of transducer deterioration.

In this project, our aim is to assess the safety of using a non-focused ultrasound device, the General Electric VIVID S70 clinical device (CE mark G1 023782 0112 ), to perform BBB ruptures in patients suffering from AD, combined with the administration of etanercept, whose bioavailability would thus be improved.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of Alzheimer's disease according to IWG2 criteria
* Biological profile in favour of Alzheimer's disease
* Age ≥ 50 years and ≤ 85 years
* Affiliated or beneficiary of a social insurance scheme
* Patient suffering from mild AD with little or no impact on autonomy, MMSE score ≥20 at inclusion
* Fazekas score <=1
* Presence of a family or a person at home who can monitor the occurrence of adverse events
* Sufficient command of the French language to take neuropsychological tests.
* Have undergone a full neuropsychological assessment within 6 months.
* If anticholinesterase treatment, stability of treatment for at least three months.
* Signed, free and informed consent from the patient and the trusted support person.

Exclusion Criteria:

* Patient previously treated with anti-TNF alpha (e.g. etanercept).
* Other cause of major neurocognitive disorder.
* Participation in another drug study
* Absolute contraindication to MRI (e.g. pacemaker, implantable stimulator, intra-orbital metallic foreign body);
* Contraindication to lumbar puncture.
* History of bleeding diathesis;
* Severe chronic respiratory disease;
* Patient on anticoagulant therapy
* Right-to-left shunt, severe pulmonary arterial hypertension;
* Known cerebral vasculopathy; (Fazekas greater than 1), sequelae of ACI.
* Treatment with Anakinra, abatacept or sulfasalazine.
* Patients who have undergone major surgery within 28 days of the first day of the study.
* Allergy to gadolinium, or any contraindication to contrast products used for brain imaging (in particular severe renal insufficiency with a glomerular filtration rate <30 ml / min / 1.73 m2).
* Allergy to xylocaine
* Epilepsy or drugs that lower the epileptogenic threshold (see Appendix 6).
* Major depressive syndrome despite appropriate treatment and/or psychotic symptoms (according to DSM IV);
* MRI characteristic of an active or acute neurological process (infection, tumour) or macro-haemorrhage.
* Non-menopausal women
* Patient benefiting from a legal protection measure other than guardianship or curatorship.
* Optic neuritis
* Manifestations of multiple sclerosis
* Live vaccinations (yellow fever, BCG) within 4 weeks of starting etanercept treatment.
* History of hepatitis B or C
* Patients with recent acute coronary syndrome or unstable ischaemic heart disease.
* History of recurrent or chronic infections, or a predisposing condition such as severe or poorly controlled diabetes.
* Patients who have undergone major surgery within 28 days of the first day of the study.

Contraindications related to etanercept :

* Hypersensitivity to etanercept or to any of the excipients of Benepali
* Sepsis or risk of sepsis
* Active infection including chronic or localised infections.

Contraindications associated with SonoVue (ultrasound contrast medium)

* Hypersensitivity to Sonovue.
* Right-to-left shunt
* Severe PAH (pulmonary arterial pressure greater than 90 mmHg)
* Uncontrolled hypertension
* Respiratory distress syndrome
* Conditions suggesting cardiovascular instability for which dobutamine is contraindicated

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of a strategy combining 9 weeks of etanercept administration with 5 weeks of repeated contrast ultrasound of 2 sessions per day, 5 days per week (from the fifth week of etanercept treatment) in patients with Alzheimer's disease. | from Day1 of repeated contrast ultrasound to Month 3 after the end of repeated contrast ultrasound
  Number of patients presenting related adverse events (CTCAE v4.0)

IPD SHARING:
Plan to Share IPD: No